CLINICAL TRIAL: NCT01405222
Title: Objective Measure of COPD Exacerbation Using the Hull Automated Cough Recorder. Verifying Use of Automated Recording Systems in Measuring Symptoms Associated With a COPD Exacerbation
Brief Title: Cough Frequency in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: 25042011
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: COPD Exacerbation
Keywords: exacerbation; COPD; Cough
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute COPD exacerbation: Patients admitted in to hospital with an acute exacerbation of COPD

SUMMARY:
Acute exacerbations of COPD remain a common cause of morbidity and are associated with a sustained increase in the normal respiratory symptoms of dyspnoea, cough, and sputum volume and purulence. It has previously been shown that a change in cough symptoms occurs in 51.7% of exacerbations in COPD. We wish to record cough during a COPD exacerbation to determine whether this can be a objective marker of exacerbation duration and severity.

DETAILED DESCRIPTION:
Acute exacerbations of COPD remain a common cause of morbidity and are associated with a sustained increase in the respiratory symptoms of dyspnoea, cough, sputum volume and sputum purulence. Cough is one of the most commonly reported and key symptoms in COPD patients. Cough can also be a useful factor in finding patients at risk of progressive airflow obstruction and cough along with the breathlessness is the major cause of distress in patients with chronic obstructive airways disease (COPD). There is limited literature looking into cough and COPD especially objective assessments.

in clinical practice and in most clinical trials scoring systems ie quality of life questionnaires or visual analogue scores, have been used to measure COPD exacerbation severity, although these may give an indication of the perceived severity of the symptom, they are inherently subjective and may be influenced by other factors. Shortfalls have prompted the development of cough recorders as an objective measure of this symptom. With this in mind we propose recruit 30 subjects with non-infective exacerbations of COPD and monitor their cough frequency as an inpatient in acute exacerbation and for 45 days post hospital discharge in order to elucidate the natural history of cough during and after an exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Male/females aged between 40-80 years.
* Previous diagnosis of COPD.
* Acute exacerbation of COPD requiring treatment with antibiotics and/or corticosteroids.
* Symptoms of increased breathlessness, cough, sputum volume or sputum purulence.
* Acute exacerbation of COPD hospitalised within 48 hrs of study participation.
* On a stable therapeutic regimen for COPD for 8 weeks prior to inclusion.
* Known history of cigarette smoking at least 10 pack yrs.
* Willing and able to comply with study procedures.
* Able to provide written informed consent to participate.

Exclusion Criteria:

* Acute exacerbation of COPD within 8 weeks prior to inclusion.
* Clinically significant or unstable concurrent disease e.g. left ventricular failure, diabetes mellitus.
* On long-term oxygen therapy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital admissions
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in recorded cough counts/hr | 5 days
  The primary objective is to evaluate the effectiveness of Hull Automated Cough Counter in recording transition of an acute COPD exacerbation. Change in no coughs/hr will be measured between start of exacerbation (day 0) to day 5 of exacerbation

SECONDARY OUTCOMES:
compare cough/hr measured via Hull automated cough counter with that of Phillips 45 day cough monitor | 45 days
  The Key secondary endpoint will be to validate automated cough counts measured via the HACC with those measured via the Phillips 45CM at day 1, 5, 20 and 45. Cough monitor results will be compared using a bland altman plot, to determine if the systems are comparative with on another

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, MD, MPhil, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Redspiratory medicine, Clinical trials Unit, Castle Hill hospital, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Result] Crooks MG, den Brinker A, Hayman Y, Williamson JD, Innes A, Wright CE, Hill P, Morice AH. Continuous Cough Monitoring Using Ambient Sound Recording During Convalescence from a COPD Exacerbation. Lung. 2017 Jun;195(3):289-294. doi: 10.1007/s00408-017-9996-2. Epub 2017 Mar 28. PMID 28353117
- See also: Publication Link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5437191/